CLINICAL TRIAL: NCT04361890
Title: Validity of Ultrasound in Women Having Pelvic Floor Muscle Training
Brief Title: Ultrasound and Pelvic Floor Muscle Training
Acronym: ERP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A01425-52
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Urinary Incontinence,Stress; Ultrasound; Elastography; Contraction; Pelvic; Urethral Hypermobility
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: ultrasonographic measurements before and after pelvic floor muscle training
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with predominant SUI (Other): All women with predominant SUI will be referred to a physiotherapist for PFMT as usually. They will have an ultrasound evaluation before and after the session
  Interventions: Diagnostic Test: perineal ultrasound

INTERVENTIONS:
Diagnostic Test: perineal ultrasound — all women will have ultrasound measurements of the bladder neck descent, of the movement of the ano-rectal angle during a Valsalva maneuver and elastographic measurement before and after PFMT. All measurement will be conducted by perineal route, with is a non invasive ultrasound route

SUMMARY:
The objective is to validate the use of ultrasound measurements (urethral mobility, movement of the ano-rectal angle, elastography measurements) in women with urinary incontiennce before and after pelvic floor muscle training (PFMT) : inter and intra-observer reproducibility; correlation with clinical examination (modified Oxford scale); sensitivity to change before/after pelvic floor muscle training

DETAILED DESCRIPTION:
Introduction: Stress urinary incontinence (SUI) is defined by involuntary loss of urine. According to the literature, its prevalence ranges from 30 to 60%. The first-line treatment of SUI is pelvic floor muscle training (PFMT). The assessment of pelvic floor muscle (PFM) contraction is essentially clinical, based on the modified OXFORD system associated with symptom questionnaires. Ultrasound is more widely used in case of SUI but has never been evaluated before and after PFMT.

Objective: The main objective of this study will be to carry out a validation study of ultrasound measurements in women with predominant SUI (urethral mobility, movement of the ano-rectal angle, elastography): Inter/intra-observer reproducibility; variability versus measurement by correlation with clinical examination (modified Oxford scale); sensitivity to change before/after PFMT Secondary objectives will be to show a correlation between the different ultrasound measurements and the clinical symptoms assessed by validated questionnaires : International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) and Contilife. A quantitative pulseal elastography analysis by Ultra-fast shear wave elastography (Supersonic Imagine) will also be performed before and after PFMT, looking for changes after PFMT. We Patient satisfaction after PFMT will also be assessed using the validated "Patient Global Impression of Improvement" questionnaire (PGI-I) Materials and Methods: This is a single-center prospective study involving patients in PFMT for predominant SUI. Patients will have a 10-week PFMT protocol. An evaluation will be conducted at the beginning and end of the program. This will include an assessment of symptoms using validated questionnaires (ICIQ-SF, CONTILIFE), a clinical examination (modified Oxford scale), as well as transperineal ultrasound measurements of urethral mobility (Bladder Neck Desent, BND measured in centimeters), movement of ano-rectal angle and quantitative elastography measurements (Ultra-fast shear wave, elasticity E expressed in kiloP).

ELIGIBILITY:
Inclusion Criteria:

* women over 18 years old
* referred for predominant SUI
* agreeing to participate in the study
* beneficiary of a social security scheme or entitled
* having been informed about the study (non-opposition)

Exclusion Criteria:

* Minor patients, under guardianship, under curator
* Patients who do not understand French
* Pregnant women
* Women with stage 2 or more prolapse according to the POP-Q classification
* Women with a history of:
* pelvis / spine trauma
* perineal pain
* urinary or vaginal infection
* perineal surgery for urinary incontinence and/or prolapse
* spinal surgery
* pacemaker
* respiratory pathology
* neurological disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Bladder neck descent reliability before PFMT | 2 years
  2 measurements of the bladder neck descent during a Valsalva maneuver (as described by Dietz et al.) will be conducted by two operators using perineal ultrasound
ano-rectal angle mobility reliability before PFMT | 2 years
  2 measurements of the ano-rectal angle mobility during a Valsalva maneuver will be conducted by two operators using perineal ultrasound
perineal elastography reliability before PFMT | 2 years
  2 measurements of perineal elastography (periurethral measurements) will be conducted by two operators using perineal ultrasound
bladder neck descent change after PFMT | 2 years
  comparison of the bladder neck descent during a Valsalva maneuver (as described by Dietz et al.) will be conducted before and after PFMT using perineal ultrasound
ano-rectal angle mobility change after PFMT | 2 years
  comparison of the ano-rectal angle mobility during a Valsalva maneuver will be conducted before and after PFMT using perineal ultrasound
perineal elastogaphy change after PFMT | 2 years
  comparison of perineal elastography (periurethral measurements) will be conducted before and after PFMT using perineal ultrasound

SECONDARY OUTCOMES:
correlation analyses between bladder neck descent measurements and urinary symptoms | 2 years
  the bladder neck descent measurements will be compared before and after PFMT to the urinary symptoms using the validated questionnaire ICIQ-SF (International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form)
patients satisfaction after pelvic floor muscle training | 2 years
  the satisfaction will be assessed using the validated questionnaire "Patient Global Impression of Improvement" (PGI-I) after PFMT

CONTACTS AND LOCATIONS:
Overall Officials: Clemence Tomadesso, PhD, Study Chair — University Hospital of Caen
Locations (1):
- Pizzoferato, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] DeLancey JO. Structural support of the urethra as it relates to stress urinary incontinence: the hammock hypothesis. Am J Obstet Gynecol. 1994 Jun;170(6):1713-20; discussion 1720-3. doi: 10.1016/s0002-9378(94)70346-9. PMID 8203431
- [Background] Petros PE, Ulmsten UI. An integral theory and its method for the diagnosis and management of female urinary incontinence. Scand J Urol Nephrol Suppl. 1993;153:1-93. No abstract available. PMID 8108659
- [Background] Fritel X, Fauconnier A, Bader G, Cosson M, Debodinance P, Deffieux X, Denys P, Dompeyre P, Faltin D, Fatton B, Haab F, Hermieux JF, Kerdraon J, Mares P, Mellier G, Michel-Laaengh N, Nadeau C, Robain G, de Tayrac R, Jacquetin B; French College of Gynaecologists and Obstetricians. Diagnosis and management of adult female stress urinary incontinence: guidelines for clinical practice from the French College of Gynaecologists and Obstetricians. Eur J Obstet Gynecol Reprod Biol. 2010 Jul;151(1):14-9. doi: 10.1016/j.ejogrb.2010.02.041. Epub 2010 Mar 16. PMID 20236751
- [Background] Hermieu JF, Denys P, Fritel X. [Critical review of guidelines for female urinary incontinence diagnosis and treatment]. Prog Urol. 2012 Oct;22(11):636-43. doi: 10.1016/j.purol.2012.08.004. Epub 2012 Sep 10. French. PMID 22999088
- [Background] Messelink B, Benson T, Berghmans B, Bo K, Corcos J, Fowler C, Laycock J, Lim PH, van Lunsen R, a Nijeholt GL, Pemberton J, Wang A, Watier A, Van Kerrebroeck P. Standardization of terminology of pelvic floor muscle function and dysfunction: report from the pelvic floor clinical assessment group of the International Continence Society. Neurourol Urodyn. 2005;24(4):374-80. doi: 10.1002/nau.20144. No abstract available. PMID 15977259
- [Background] Deffieux X, Billecocq S, Demoulin G, Rivain AL, Trichot C, Thubert T. [Pelvic floor rehabilitation for female urinary incontinence: mechanisms of action]. Prog Urol. 2013 Jun;23(8):491-501. doi: 10.1016/j.purol.2013.04.002. Epub 2013 May 2. French. PMID 23725579
- [Background] Miller JM, Sampselle C, Ashton-Miller J, Hong GR, DeLancey JO. Clarification and confirmation of the Knack maneuver: the effect of volitional pelvic floor muscle contraction to preempt expected stress incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jun;19(6):773-82. doi: 10.1007/s00192-007-0525-3. PMID 18204797
- [Background] Hung HC, Hsiao SM, Chih SY, Lin HH, Tsauo JY. Effect of pelvic-floor muscle strengthening on bladder neck mobility: a clinical trial. Phys Ther. 2011 Jul;91(7):1030-8. doi: 10.2522/ptj.20100186. Epub 2011 May 12. PMID 21566065
- [Background] Schaer GN, Perucchini D, Munz E, Peschers U, Koechli OR, Delancey JO. Sonographic evaluation of the bladder neck in continent and stress-incontinent women. Obstet Gynecol. 1999 Mar;93(3):412-6. doi: 10.1016/s0029-7844(98)00420-7. PMID 10074990
- [Background] Balmforth JR, Mantle J, Bidmead J, Cardozo L. A prospective observational trial of pelvic floor muscle training for female stress urinary incontinence. BJU Int. 2006 Oct;98(4):811-7. doi: 10.1111/j.1464-410X.2006.06393.x. PMID 16978276
- [Background] Tosun OC, Solmaz U, Ekin A, Tosun G, Gezer C, Ergenoglu AM, Yeniel AO, Mat E, Malkoc M, Askar N. Assessment of the effect of pelvic floor exercises on pelvic floor muscle strength using ultrasonography in patients with urinary incontinence: a prospective randomized controlled trial. J Phys Ther Sci. 2016 Jan;28(2):360-5. doi: 10.1589/jpts.28.360. Epub 2016 Feb 29. PMID 27065519
- [Background] Volloyhaug I, Morkved S, Salvesen O, Salvesen KA. Assessment of pelvic floor muscle contraction with palpation, perineometry and transperineal ultrasound: a cross-sectional study. Ultrasound Obstet Gynecol. 2016 Jun;47(6):768-73. doi: 10.1002/uog.15731. Epub 2016 May 2. PMID 26300128
- [Background] Dietz HP. Ultrasound imaging of the pelvic floor. Part I: two-dimensional aspects. Ultrasound Obstet Gynecol. 2004 Jan;23(1):80-92. doi: 10.1002/uog.939. PMID 14971006
- [Background] Bergman A, McKenzie CJ, Richmond J, Ballard CA, Platt LD. Transrectal ultrasound versus cystography in the evaluation of anatomical stress urinary incontinence. Br J Urol. 1988 Sep;62(3):228-34. doi: 10.1111/j.1464-410x.1988.tb04324.x. PMID 3056562
- [Background] Johnson JD, Lamensdorf H, Hollander IN, Thurman AE. Use of transvaginal endosonography in the evaluation of women with stress urinary incontinence. J Urol. 1992 Feb;147(2):421-5. doi: 10.1016/s0022-5347(17)37256-7. PMID 1732608
- [Background] Wise BG, Burton G, Cutner A, Cardozo LD. Effect of vaginal ultrasound probe on lower urinary tract function. Br J Urol. 1992 Jul;70(1):12-6. doi: 10.1111/j.1464-410x.1992.tb15655.x. PMID 1638367
- [Background] Alper T, Cetinkaya M, Okutgen S, Kokcu A, Malatyalioglu E. Evaluation of urethrovesical angle by ultrasound in women with and without urinary stress incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(5):308-11. doi: 10.1007/s001920170031. PMID 11715996
- [Background] Koelbl H, Bernaschek G. A new method for sonographic urethrocystography and simultaneous pressure-flow measurements. Obstet Gynecol. 1989 Sep;74(3 Pt 1):417-22. PMID 2668819
- [Background] Thompson JA, O'Sullivan PB, Briffa K, Neumann P, Court S. Assessment of pelvic floor movement using transabdominal and transperineal ultrasound. Int Urogynecol J Pelvic Floor Dysfunct. 2005 Jul-Aug;16(4):285-92. doi: 10.1007/s00192-005-1308-3. Epub 2005 Mar 22. PMID 15782286
- [Background] Dietz HP, Clarke B, Herbison P. Bladder neck mobility and urethral closure pressure as predictors of genuine stress incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2002;13(5):289-93. doi: 10.1007/s001920200063. PMID 12355287
- [Background] Dietz HP, Clarke B. The influence of posture on perineal ultrasound imaging parameters. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(2):104-6. doi: 10.1007/pl00004030. PMID 11374506
- [Background] Yang SH, Huang WC, Yang SY, Yang E, Yang JM. Validation of new ultrasound parameters for quantifying pelvic floor muscle contraction. Ultrasound Obstet Gynecol. 2009 Apr;33(4):465-71. doi: 10.1002/uog.6338. PMID 19306473
- [Background] Ferraioli G, Tinelli C, Zicchetti M, Above E, Poma G, Di Gregorio M, Filice C. Reproducibility of real-time shear wave elastography in the evaluation of liver elasticity. Eur J Radiol. 2012 Nov;81(11):3102-6. doi: 10.1016/j.ejrad.2012.05.030. Epub 2012 Jun 27. PMID 22749107
- [Background] Berg WA, Cosgrove DO, Dore CJ, Schafer FK, Svensson WE, Hooley RJ, Ohlinger R, Mendelson EB, Balu-Maestro C, Locatelli M, Tourasse C, Cavanaugh BC, Juhan V, Stavros AT, Tardivon A, Gay J, Henry JP, Cohen-Bacrie C; BE1 Investigators. Shear-wave elastography improves the specificity of breast US: the BE1 multinational study of 939 masses. Radiology. 2012 Feb;262(2):435-49. doi: 10.1148/radiol.11110640. PMID 22282182
- [Background] Cosgrove DO, Berg WA, Dore CJ, Skyba DM, Henry JP, Gay J, Cohen-Bacrie C; BE1 Study Group. Shear wave elastography for breast masses is highly reproducible. Eur Radiol. 2012 May;22(5):1023-32. doi: 10.1007/s00330-011-2340-y. Epub 2011 Dec 31. PMID 22210408
- [Background] Aljuraifani R, Stafford RE, Hug F, Hodges PW. Female striated urogenital sphincter contraction measured by shear wave elastography during pelvic floor muscle activation: Proof of concept and validation. Neurourol Urodyn. 2018 Jan;37(1):206-212. doi: 10.1002/nau.23275. Epub 2017 Apr 13. PMID 28407305
- [Background] Stafford RE, Aljuraifani R, Hug F, Hodges PW. Application of shear-wave elastography to estimate the stiffness of the male striated urethral sphincter during voluntary contractions. BJU Int. 2017 Apr;119(4):619-625. doi: 10.1111/bju.13688. Epub 2016 Nov 11. PMID 27753239
- [Background] Kreutzkamp JM, Schafer SD, Amler S, Strube F, Kiesel L, Schmitz R. Strain Elastography as a New Method for Assessing Pelvic Floor Biomechanics. Ultrasound Med Biol. 2017 Apr;43(4):868-872. doi: 10.1016/j.ultrasmedbio.2016.12.004. Epub 2017 Jan 17. PMID 28108041
- [Background] Pizzoferrato AC, Fauconnier A, Bader G. [Value of ultrasonographic measurement of bladder neck mobility in the management of female stress urinary incontinence]. Gynecol Obstet Fertil. 2011 Jan;39(1):42-8. doi: 10.1016/j.gyobfe.2010.09.019. Epub 2010 Dec 24. French. PMID 21185762
- [Background] Srikrishna S, Robinson D, Cardozo L. Validation of the Patient Global Impression of Improvement (PGI-I) for urogenital prolapse. Int Urogynecol J. 2010 May;21(5):523-8. doi: 10.1007/s00192-009-1069-5. Epub 2009 Dec 15. PMID 20013110
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Amarenco G, Arnould B, Carita P, Haab F, Labat JJ, Richard F. European psychometric validation of the CONTILIFE: a Quality of Life questionnaire for urinary incontinence. Eur Urol. 2003 Apr;43(4):391-404. doi: 10.1016/s0302-2838(03)00054-x. PMID 12667721